CLINICAL TRIAL: NCT05405998
Title: Development of a Proactive Health Care Pathway When Initiating Continuous Subcutaneous Apomorphine Infusion in Patients With Parkinson Disease : Impact on Their Autonomy
Brief Title: Development of a Proactive Health Care Pathway When Initiating Continuous Subcutaneous Apomorphine Infusion in Patients With Parkinson Disease : Impact on Their Autonomy (AUTAP)
Acronym: AUTAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-A01424-37
Record Dates: First submitted 2022-05-17; First posted 2022-06-06 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group : proactive course (Experimental): The strategy is based on the implementation of an "optimized" proactive care pathway, combining elements that promote city-hospital coordination in setting up the pump and elements that promote patient education.
  Interventions: Other: Proactive care pathway
- Control group : optimized medical treatment (No Intervention): At the end of the inclusion visit (see previous chapter), the patient will be invited to come to the hospital two weeks later for pump placement.

INTERVENTIONS:
Other: Proactive care pathway — Patient participation in a specific therapeutic education program, as soon as the therapeutic decision is made.
  The reinforced cooperation of the expert centers with the homecare providers on 2 different times:
  1. before the installation of the pump, i.e. before the episode of hospitalization dedicated to the starting of the treatment;
  2. after the installation of the pump following the above mentioned hospitalization.
  Arms: Experimental group : proactive course

SUMMARY:
Continuous subcutaneous apomorphine infusion (CSAI) has proven to be effective in advaced Parkinson's disease patients with motor fluctuations not controlled by oral or transdermal medication. After initiation of this therapy, most of the patients need nurse services at home for the entire duration of treatment. Some patients are reluctant about this dependence and thus may refuse or delay the initiation of CSAI. To date, there is no guideline to promote patients' autonomy in managing CSAI treatment. Thus we developed a program focusing on early autonomy during CSAI intitiation, through empowering the patient or their carer, and promoting primary and tertiary care.

The hypothesis is that implementing the program will lead patients to autonomy. This will have beneficial effects on clinical and heath-related outcomes and may be cost-effective.

DETAILED DESCRIPTION:
The main objective of the project is to evaluate the impact of the proactive care pathway during the installation of an apomorphine pump on the autonomy at 6 months of patients with Parkinson's disease at the stage of motor complications.

This care pathway corresponds to a care program combining therapeutic education of the patient, modification of the hospital course and city-hospital coordination. The content of this program is detailed below in chapter III.3. Experimental group: proactive care pathway.

The interest of the protocol will be evaluated at several levels: from the patients' point of view, from the caregivers' point of view, from the medico-economic point of view. Among all the indicators, the achievement of autonomy is retained as the main criterion (see chapter on main evaluation criterion).

Secondary objectives are to measure the value of the proactive care pathway on:

* Patient-related parameters Psychobehavioral factors (quality of life, self-esteem, mood...) ; Treatment persistence; Patient satisfaction; Clinical symptomatology (overall clinical impression, motor and non-motor symptoms, impulse control disorders).
* Caregiver burden.
* Use of the care system in both groups and medico-economic impact of the intervention (cost-consequence analysis and cost-utility analysis) from a societal perspective;

For this study, patients will be accompanied by their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age;
* Affiliated to the social security;
* Parkinson's disease according to the diagnostic criteria of the UK Parkinson's disease society brain bank clinical diagnostic criteria;
* Presence of disabling motor fluctuations and/or dyskinesia despite optimized oral treatment (MDS-UPDRS IV item >2)
* Patient eligible for and accepting apomorphine pump therapy
* Autonomous patient (Hoehn and Yahr stage < 4);
* No significant cognitive impairment (MoCA >= 25)
* Patient can be autonomous on the daily management of the pump according to the investigator's opinion.
* Patient having signed an informed consent

Exclusion Criteria:

* Significant cognitive impairment (MoCA score <25);
* Major depressive episode, uncontrolled at the time of assessment (BDI>25) or bipolar disorder;
* Active visual hallucinations or history of severe hallucination episodes;
* Previous apomorphine pump use;
* History of respiratory distress;
* History of severe impulse control disorders;
* Patient and/or caregiver who cannot be empowered in the opinion of the investigator.
* Protected persons, curators, persons under court protection, persons deprived of liberty by judicial or administrative decision, persons under forced psychiatric care and persons admitted to a health or social institution for purposes other than those of the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of autonomy | 6 months
  The patient will be considered autonomous if he/she does not need nursing care to manage his/her treatment and the pump for 15 days
Unified Parkinson's disease rating scale (MDS-UPDRS), section VI (Schwab and England) | 6 months
  Gold standard in the evaluation of activity in daily living in PD patients. The score varies per question from 0 to 4. If the patient scores 0, it means that he/she does not have any particular problem related to the disease. On the contrary, if the patient obtains a score of 4 for a question, it means that the disease has a severe impact on his daily life.

SECONDARY OUTCOMES:
Parkinson disease questionnaire 39 (PDQ39) | 6 months and 12 months
  Self-assessment questionnaire integrating 39 items evaluating quality of life of PD patients. Establish a score between 0 and 100.
MDS-UPDRS section II | 6 months and 12 months
  This section evaluate the motor aspects of experiences in daily living. The score varies per question from 0 to 4. If the patient scores 0, it means that he/she does not have any particular problem related to the disease. On the contrary, if the patient obtains a score of 4 for a question, it means that the disease has a severe impact on his daily life.
MDS-UPDRS section I | 6 months and 12 months
  This section evaluate the non-motor aspects of experiences of daily living.The score varies per question from 0 to 4. If the patient scores 0, it means that he/she does not have any particular problem related to the disease. On the contrary, if the patient obtains a score of 4 for a question, it means that the disease has a severe impact on his daily life.
Clinical Global impression | 6 months and 12 months
  Measured by the patient, the caregiver and the investigator. There are 2 components to the CGI (20): (i) the CGI-severity to assign a disease severity score from 1 to 7 (1=no disease; 7=very severe). (ii) the CGI-Improvement which establishes a score of improvement since the beginning of treatment between 1 and 7 (1=great improvement; 7=great deterioration)
MDS-UPDRS III and IV | 6 months and 12 months
  This section evaluate the motor examination (III) and motor complications (IV).The score varies per question from 0 to 4. If the patient scores 0, it means that he/she does not have any particular problem related to the disease. On the contrary, if the patient obtains a score of 4 for a question, it means that the disease has a severe impact on his daily life.
QUIP RS | 6 months and 12 months
  Questionnaire for impulsive-compulsive disorders in Parkinson's disease-rating scale. The score per question varies from 0 to 4. If the patient obtains a 0, it means that he/she does not have an impulse control disorder. On the contrary, if the patient gets a 4 it means that he/she has an impulse control disorder very often. The total score of the questionnaire varies between 0 and 112.
ZARIT score | 6 months and 12 months
  Assessment of caregiver burden. The score varies between 0 and 88. Score < 20: mild "burden 21 < score < 40: mild to moderate "burden 41 < score < 60 : moderate to severe "burden 61 < score < 88 : severe "burden

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- AP-HM, Marseille, France